CLINICAL TRIAL: NCT02219048
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP STUDY TO ASSESS THE EFFICACY, SAFETY, AND TOLERABILITY OF PF-03715455 ADMINISTERED TWICE DAILY BY INHALATION FOR 12 WEEKS IN SUBJECTS WITH PERSISTENT MODERATE TO SEVERE ASTHMA WHO REMAIN UNCONTROLLED DESPITE TREATMENT WITH INHALED CORTICOSTEROIDS (ICS) AND LONG-ACTING BETA2 AGONISTS (LABA)
Brief Title: An Evaluation Of PF-03715455 In Moderate To Severe Uncontrolled Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The termination was due to business reasons. No safety or efficacy concerns contributed to the termination of the study
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A9111007; INHALED P38I ASTHMA (Other: Alias Study Number)
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: Asthma; Staged withdrawal of background therapy
MeSH Terms: conditions — Asthma | interventions — N-(1-(3-chloro-4-hydroxyphenyl)-3-(1,1-dimethylethyl)-1H-pyrazol-5-yl)-N'-((2-((3-(2-((2-hydroxyethyl)thio)phenyl)-1,2,4-triazolo(4,3-a)pyridin-6-yl)thio)phenyl)methyl)-urea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matched blinded placebo
  Interventions: Drug: Placebo
- PF-03715455 (Experimental): PF-03715455
  Interventions: Drug: PF-03715455

INTERVENTIONS:
Drug: Placebo — 680 micrograms BID, Orally inhaled placebo for 12 weeks
  Arms: Placebo
Drug: PF-03715455 — 680 micrograms BID, Orally inhaled PF-03715455 for 12 weeks
  Arms: PF-03715455

SUMMARY:
The study proposes to evaluate the safety and efficacy of PF-03715455 in moderate to severe asthma when added to standard of care and during staged withdrawal of background therapy.

DETAILED DESCRIPTION:
Study terminated on 7th April 2015. The termination was due to business reasons. No safety or efficacy concerns contributed to the termination of the study

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a physician documented history or diagnosis of persistent asthma (according to GINA, 2014 definition of asthma),
* Pre bronchodilator FEV1 of greater than or equal to 50 and less that 80% of predicted.
* Subjects defined as GINA Step 4 on a stable dose of either fluticasone/salmeterol combination therapy, or budesonide/formoterol combination therapy or mometasone/formoterol combination therapy.
* Subjects who are defined as uncontrolled as evidenced by; Juniper Asthma Control Questionnaire (5 item version, ACQ) score greater than or equal to 1.5 and less than or equal to 3.0)

Exclusion Criteria:

* Subjects diagnosed with chronic pulmonary disease (COPD) and/or other chronic pulmonary diseases (eg, Occupational asthma, pulmonary fibrosis, bronchiectasis, Allergic bronchopulmonary aspergillosis (ABPA), pneumoconiosis, sarcoidosis, tuberculosis).
* Subjects who are current smokers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (28):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Pulmonary Associates, Pa, Phoenix, Arizona
  - Little Rock Allergy & Asthma Clinical Research Center, Little Rock, Arkansas
  - California Research Medical Group, Inc, Fullerton, California
  - California Allergy and Asthma Medical Group, Inc., Los Angeles, California
  - Jonathan Corren MD, Inc., Los Angeles, California
  - Integrated Research Group, Incorporated, Riverside, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Allergy Associates Medical Group, San Diego, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, PC, Denver, Colorado
  - University of South Florida - Asthma, Allergy and Immunology Clinical Research Unit, Tampa, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Chesapeake Clinical Research, Inc., Baltimore, Maryland
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Associated Specialists in Medicine, PC, St Louis, Missouri
  - The Clinical Research Center, L.L.C., St Louis, Missouri
  - The Asthma and Allergy Center, Bellevue, Nebraska
  - North Shore Long Island Jewish Health System, New Hyde Park, New York
  - American Health Research, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - University of Pittsburgh Asthma Institute, Pittsburgh, Pennsylvania
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - The Allergy & Asthma Clinic of Central Texas, Killeen, Texas
  - University of Wisconsin School of Medicine & Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9111007&StudyName=An%20Evaluation%20Of%20PF-03715455%20In%20Moderate%20To%20Severe%20Uncontrolled%20Asthma

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Twice Daily: Participants received placebo-matched PF-03715455 twice a day for 12 weeks via oral inhalation using the Miat monodose inhaler.
- PF-03715455 680 mcg Twice Daily: Participants received PF-03715455 680 micrograms (mcg) twice a day for 12 weeks via oral inhalation using the Miat monodose inhaler.
Period: Overall Study
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Started | 26 | 25
Completed | 5 | 4
Not Completed | 21 | 21
Not completed — Adverse Event | 2 | 5
Not completed — No longer meets eligibility criteria | 1 | 0
Not completed — Study terminated by sponsor | 16 | 15
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all randomized participants who received at least 1 dose of PF-03715455 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (14.1) | 44.2 (10.0) | 43.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Asthma Worsening Events
Description: Asthma worsening was defined as one of the following events: greater than or equal to (>=) 30% reduction from baseline in morning peak expiratory flow (PEF) on 2 consecutive days; >=6 additional rescue puffs of albuterol or levalbuterol in a 24-hour period (compared to baseline) on 2 consecutive days; deterioration of asthma (as determined by the Investigator) requiring systemic steroid treatment, an increase in inhaled corticosteroids >=4 times the last dose received prior to discontinuation from the study, or hospitalization due to asthma.
Time Frame: Baseline up to follow-up period (Week 16)
Population: The modified intent-to-treat (mITT) analysis set included all randomized participants who received at least 1 dose of PF-03715455 or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 26 | 25
percentage of participants | 11.5 | 16.0

2. Secondary Outcome: Time to Asthma Worsening Event
Description: The time post randomization that the first asthma worsening event occurred (defined above).
Time Frame: Baseline up to follow-up period (Week 16)
Population: The modified intent-to-treat (mITT) analysis set initially included all randomized participants who received at least 1 dose of PF-03715455 or placebo. Only 7 participants (4 in PF-03715455 and 3 in placebo) were included in the presented descriptive analysis, since other observations were censored by study termination.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 3 | 4
days | 58 [35 to 82] | 19.5 [2 to 84]

3. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Baseline was defined as the latest measurement before first dosing.
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: The mITT analysis set included all randomized participants who received at least 1 dose of PF-03715455 or placebo; n=number of participants analyzed in respective arms for category.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 26 | 25
liters
  Baseline | 2.084 (0.4645) | 2.158 (0.4917)
  Change From Baseline at Week 1 | 0.188 (0.3941) | 0.111 (0.2226)
  Change From Baseline at Week 2: number analyzed (Participants) | 23 | 23
  Change From Baseline at Week 2 | 0.244 (0.3797) | 0.107 (0.1959)
  Change From Baseline at Week 3: number analyzed (Participants) | 21 | 20
  Change From Baseline at Week 3 | 0.273 (0.3444) | 0.124 (0.2140)
  Change From Baseline at Week 4: number analyzed (Participants) | 21 | 21
  Change From Baseline at Week 4 | 0.234 (0.3251) | 0.148 (0.2217)
Statistical Analysis 1: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Change From Baseline at Week 1; Test type: Superiority or Other; Longitudinal Analysis of Covariance; LANCOVA model contained fixed factors of treatment, week, treatment/baseline by week interaction, baseline value, and unstructured covariance matrix; Mean Difference (Net) = -0.0719, 90% CI 2-sided [-0.2243 to 0.0805], Standard Error of Mean 0.0909
Statistical Analysis 2: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Change From Baseline at Week 2; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = -0.0920, 90% CI 2-sided [-0.2362 to 0.0523], Standard Error of Mean 0.0860
Statistical Analysis 3: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Change From Baseline at Week 3; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = -0.1131, 90% CI 2-sided [-0.2536 to 0.0274], Standard Error of Mean 0.0837
Statistical Analysis 4: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Change From Baseline at Week 4; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = -0.0580, 90% CI 2-sided [-0.1971 to 0.0812], Standard Error of Mean 0.0829
Statistical Analysis 5: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Change From Baseline Over Week 1 to 4; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Median Difference (Net) = -0.0837, 90% CI 2-sided [-0.2081 to 0.0406], Standard Error of Mean 0.0742

4. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 26 | 25
liters
  Baseline | 3.393 (0.8966) | 3.384 (0.8958)
  Change at Week 1 | 0.140 (0.3866) | 0.042 (0.2401)
  Change at Week 2: number analyzed (Participants) | 23 | 23
  Change at Week 2 | 0.243 (0.3813) | 0.066 (0.2321)
  Change at Week 3: number analyzed (Participants) | 21 | 20
  Change at Week 3 | 0.252 (0.3053) | 0.020 (0.2784)
  Change at Week 4: number analyzed (Participants) | 21 | 21
  Change at Week 4 | 0.178 (0.3028) | 0.080 (0.3136)

5. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 6 Seconds (FEV6)
Description: FEV6 is the maximal volume of air exhaled in the first 6 seconds of a forced expiration from a position of full inspiration.
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 26 | 25
liters
  Baseline | 3.175 (0.7707) | 3.150 (0.7546)
  Change at Week 1 | 0.134 (0.3782) | 0.078 (0.2401)
  Change at Week 2: number analyzed (Participants) | 23 | 23
  Change at Week 2 | 0.221 (0.3603) | 0.072 (0.1922)
  Change at Week 3: number analyzed (Participants) | 21 | 20
  Change at Week 3 | 0.264 (0.3149) | 0.069 (0.2569)
  Change at Week 4: number analyzed (Participants) | 21 | 21
  Change at Week 4 | 0.178 (0.2986) | 0.106 (0.2664)

6. Secondary Outcome: Change From Baseline in Asthma Symptom Scores
Description: Participants used a daily diary assessment to record overall asthma symptom scores twice a day (morning and evening). Questions included extent of albuterol use, symptoms of wheezing, breathlessness, chest tightness, and cough. The visit dependent asthma symptom scores were calculated based on the item in the daily diary assessment. A participant summarized her/his daily frequency of asthma symptoms during the last 24 hours by the assignment of an integer score (0,1,2,3 or 4). The score=0 value denoted the day without symptoms and the score=4 value denoted the day where symptoms occurred all of the time. The asthma symptom scores were calculated by averaging the values of the daily scores within visit-dependent time window. Higher score indicates asthma worsening
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 26 | 25
units on a scale
  Baseline | 1.15 (0.567) | 1.23 (0.636)
  Change at Week 1 | -0.14 (0.406) | -0.12 (0.453)
  Change at Week 2: number analyzed (Participants) | 23 | 23
  Change at Week 2 | -0.17 (0.497) | -0.36 (0.560)
  Change at Week 3: number analyzed (Participants) | 21 | 20
  Change at Week 3 | -0.15 (0.471) | -0.44 (0.458)
  Change at Week 4: number analyzed (Participants) | 21 | 21
  Change at Week 4 | -0.19 (0.565) | -0.38 (0.513)
Statistical Analysis 1: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Change From Baseline Averaged Over Week 1 to 4; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.090, 90% CI 2-sided [-0.285 to 0.106], Standard Error of Mean 0.116

7. Secondary Outcome: Number of Night Time Awakenings Per Week
Description: The number of nocturnal awakenings due to asthma symptoms was recorded by the participant.
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: night awakenings per week
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 26 | 25
night awakenings per week
  Baseline | 2.03 (2.088) | 1.40 (1.925)
  Week 1 | 1.34 (2.101) | 1.38 (2.210)
  Week 2: number analyzed (Participants) | 23 | 23
  Week 2 | 1.39 (1.990) | 1.43 (2.251)
  Week 3: number analyzed (Participants) | 21 | 20
  Week 3 | 0.89 (1.657) | 1.66 (2.431)
  Week 4: number analyzed (Participants) | 21 | 21
  Week 4 | 1.04 (1.869) | 1.27 (1.830)

8. Secondary Outcome: Change From Baseline in Morning and Evening Peak Expiratory Flow (PEF)
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. The changes from baseline (CFB) at each week and over 4 weeks were analyzed.
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 26 | 25
liters per minute
  Morning PEF: Baseline | 346.67 (92.666) | 361.46 (145.788)
  Morning PEF: CFB at Week 1 | 17.42 (31.100) | 22.25 (41.585)
  Morning PEF: CFB at Week 2: number analyzed (Participants) | 23 | 23
  Morning PEF: CFB at Week 2 | 22.25 (38.822) | 29.80 (51.818)
  Morning PEF: CFB at Week 3: number analyzed (Participants) | 21 | 20
  Morning PEF: CFB at Week 3 | 18.86 (40.775) | 23.55 (42.129)
  Morning PEF: CFB at Week 4: number analyzed (Participants) | 21 | 21
  Morning PEF: CFB at Week 4 | 21.54 (41.697) | 22.65 (47.892)
  Evening PEF: Baseline | 357.86 (91.426) | 382.05 (130.316)
  Evening PEF: CFB at Week 1 | 20.51 (33.868) | 20.14 (43.925)
  Evening PEF: CFB at Week 2: number analyzed (Participants) | 23 | 23
  Evening PEF: CFB at Week 2 | 20.70 (29.127) | 23.87 (40.435)
  Evening PEF: CFB at Week 3: number analyzed (Participants) | 21 | 20
  Evening PEF: CFB at Week 3 | 22.55 (35.234) | 17.74 (44.378)
  Evening PEF: CFB at Week 4: number analyzed (Participants) | 21 | 21
  Evening PEF: CFB at Week 4 | 19.10 (42.063) | 23.22 (48.329)
Statistical Analysis 1: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Morning PEF: CFB at Week 1; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 6.017, 90% CI 2-sided [-10.760 to 22.794], Standard Error of Mean 10.003
Statistical Analysis 2: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Morning PEF: CFB at Week 2; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 6.591, 90% CI 2-sided [-13.926 to 27.108], Standard Error of Mean 12.228
Statistical Analysis 3: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Morning PEF: CFB at Week 3; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.954, 90% CI 2-sided [-18.644 to 20.552], Standard Error of Mean 11.673
Statistical Analysis 4: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Morning PEF: CFB at Week 4; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -4.368, 90% CI 2-sided [-26.069 to 17.333], Standard Error of Mean 12.920
Statistical Analysis 5: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Morning PEF: CFB Averaged Over 4 Weeks; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 2.299, 90% CI 2-sided [-15.323 to 19.920], Standard Error of Mean 10.503
Statistical Analysis 6: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Evening PEF: CFB at Week 1; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 1.135, 90% CI 2-sided [-17.248 to 19.519], Standard Error of Mean 10.961
Statistical Analysis 7: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Evening PEF: CFB at Week 2; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 2.834, 90% CI 2-sided [-13.871 to 19.540], Standard Error of Mean 9.956
Statistical Analysis 8: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Evening PEF: CFB at Week 3; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.374, 90% CI 2-sided [-27.933 to 11.185], Standard Error of Mean 11.652
Statistical Analysis 9: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Evening PEF: CFB at Week 4; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.445, 90% CI 2-sided [-23.245 to 22.356], Standard Error of Mean 13.573
Statistical Analysis 10: Comparison: Placebo Twice Daily vs PF-03715455 680 mcg Twice Daily; Evening PEF: CFB Averaged Over 4 Weeks; Test type: Superiority or Other; Longitudinal Analysis of Covariance; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.212, 90% CI 2-sided [-18.520 to 16.096], Standard Error of Mean 10.317

9. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ)-5 Score at Week 1, Week 2, Week 3, and Week 4
Description: The 5-question version of the Juniper ACQ is a validated questionnaire to evaluate asthma control. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ score was the mean of the responses. Mean scores of <= 0.75 indicate well-controlled asthma, scores between 0.76 and less than (<) 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma.
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 26 | 25
units on a scale
  Baseline | 2.18 (0.315) | 2.17 (0.489)
  Change at Week 1 | -0.50 (0.742) | -0.27 (0.658)
  Change at Week 2: number analyzed (Participants) | 23 | 23
  Change at Week 2 | -0.66 (0.826) | -0.53 (0.670)
  Change at Week 3: number analyzed (Participants) | 21 | 20
  Change at Week 3 | -0.62 (0.959) | -0.34 (0.751)
  Change at Week 4: number analyzed (Participants) | 21 | 21
  Change at Week 4 | -0.71 (0.838) | -0.41 (0.806)

10. Secondary Outcome: Number of Daily Puffs of Rescue Medication
Description: The use of rescue bronchodilators (albuterol or levalbuterol) for symptomatic relief of asthma in a 24-hour period was recorded by the participant.
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: puffs per day
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 26 | 25
puffs per day
  Baseline | 1.90 (1.364) | 1.96 (1.628)
  Week 1 | 1.51 (1.254) | 1.74 (2.164)
  Week 2: number analyzed (Participants) | 23 | 23
  Week 2 | 1.51 (1.431) | 1.07 (1.494)
  Week 3: number analyzed (Participants) | 21 | 20
  Week 3 | 1.48 (1.391) | 1.37 (1.772)
  Week 4: number analyzed (Participants) | 21 | 21
  Week 4 | 1.34 (1.385) | 1.54 (2.264)

ADVERSE EVENTS:
Time Frame: Baseline up to 1 month after end-of-treatment visit (Week 12)
Arm/Group | Placebo Twice Daily | PF-03715455 680 mcg Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 10/26 | 15/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Twice Daily (N=26) | PF-03715455 680 mcg Twice Daily (N=25)
Dry eye (Eye disorders) | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Influenza-like illness (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Forced expiratory volume decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 1 | 0
Middle insomnia (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oral candidiasis (Infections and infestations) | 2 | 3
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
The study was terminated early due to portfolio prioritization. Most participants observations of time to asthma worsening event were censored by the study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.